# Statistical Analysis Plan

Identifiers: NCT02189213

Protocol ID: 6884

Title: Treatment of Pediatric Anxiety Disorders by Predicting Treatment Response Through Biocellular Markers and Sleep Module

PI: Amir Levine

Date: 08/30/2021

#### Introduction

## **Background**

Anxiety disorders are among the most common and debilitating psychiatric conditions in youth, affecting more than 10% of all children and adolescents. Selective-serotonin reuptake inhibitors (SSRIs)—the first-line psychopharmacologic treatment for pediatric anxiety disorders—produce benefit in only 50-60% of patients and can take up to 12 weeks to improve symptoms.

Study Design

### **METHODS**

We conducted a prospective, open-label trial of flexibly-dosed sertraline in children and adolescents with generalized, separation and or social anxiety disorders.

## Aims and Objectives

To measure improvement after treatment with sertraline using the Clinical Global Impressions Improvement (CGI-I) Scale

Hypothesis: At least 50% of subjects will respond to Sertraline treatment (CGI-I greater than or equal to 2).

#### Outcomes

# Primary outcomes

The primary outcome in the study was response to sertraline measured by the Clinical Global Impressions Improvement (CGI-I) Scale.

Response to Sertraline was defined as The Clinical Global Impressions Scale Clinical Global Impressions Improvement (CGI-I) Scale, an instrument used to quantify and track patient progress and treatment response over time.

The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.

The CGI-Improvement scale comprises a one-item measures evaluating the following change from the initiation of treatment on a seven-point scale.

The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no

change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.

CGI-I scale of 1-2 is considered response to treatment. Anything below that (3-7) is considered non-response to sertraline treatment.

# Analyses

## **RESULTS**

7 patients completed the trial. Out of the 7 three were non-responders CGI-I less than 2, and 4 were responders, CGI-I score equal to or greater than 2 two-tail t-test was performed.

# Safety outcomes

There were no serious adverse events.